CLINICAL TRIAL: NCT04185025
Title: Compare the Skin Barrier Repair Function of Two Ceramide Containing Moisturizers: A Double-blind, Randomized, Controlled Trial
Brief Title: Compare the Skin Barrier Repair Function of Two Ceramide Containing Moisturizers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Wu, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: v2.0
Record Dates: First submitted 2019-11-29; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: CeraVe Moisturising Lotion
MeSH Terms: interventions — Ceramides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CeraVe Moisturising Lotion (Experimental)
  Interventions: Drug: Ceramides
- Half Mu ceramide body milk (Active Comparator)
  Interventions: Drug: Ceramides

INTERVENTIONS:
Drug: Ceramides — On the 0th day, it is determined that one of the leg extensions of the participant is the test side using CeraVe Moisturising Lotion and the opposite side is the control side using Half Mu ceramide body milk by the random table. Participants are required to use the product in the morning and evening according to the "Product Use Procedures", during which other moisturizing products or emollients are prohibited. And the follow-up tests are conducted at the prescribed time. At each visit, empty packaging of products used during this period must be collected; if they are not used up as required, the remaining products must be collected.

SUMMARY:
This study aims to evaluate the improvement of CeraVe moisturising lotion on the cuticle moisture of dry skin and barrier repair function.

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteer to participate in the trial, sign the informed consent, be able to cooperate with follow-up observation, and conduct the trial according to the guidance of the doctor.
* Dry skin subjects with symmetrical distribution of forearm flexion diagnosed by a doctor.
* Those who are 30-80 years old, male or female.
* Those with good compliance who can not use other external drugs during the entire observation period.

Exclusion Criteria:

* Those who do not sign the informed consent.
* Those with the history of allergies to test product and control product ingredients.
* Those who received or are receiving medical or physical therapy for any skin or systemic disease recently (≤3 months)
* Those who have a large amount of exudation in the acute phase or who are infected at the test site.
* Female subjects who are preparing for pregnancy, pregnancy, lactation, or within six months after delivery.
* Those who participate in clinical trials of other moisturizing products or emollients.
* Those who are taking other oral medicines that affect the skin condition.
* Those who the investigator considers unsuitable for other reasons.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Self-assessment from patients | 17 days
  The patients fill out questionnaires and score erythema, desquamation, dryness, itching, and cleft palate on both sides of the calves (0 = none, 1 = light, 2 = medium, 3 = severe).

SECONDARY OUTCOMES:
The loss of transdermal water | 0 day, 1 day, 7 days, 14 days, 17 days
  The percutaneous water loss value of the test site is measured continuously in an open chamber with Tewameter (TM300, Courage and Khazaka, Germany), and the measurement is performed 3 times continuously. The average value is taken after the value is stable.
Cuticle moisture | 0 day, 1 day, 7 days, 14 days, 17 days
  The water content in the stratum corneum of the test site is measured 5 times with Corneometer (CM825, Course and Khazaka, Germany) and the average value is taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China